CLINICAL TRIAL: NCT03091712
Title: Insulin Degludec Titration Using Mobile Insulin Dosing System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glooko (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GL3
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Degludec; MIDS; Mobile Insulin Dosing System; Glooko; Tresiba; Tresiba® U-200 FlexTouch®
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Prospective, open label, randomized, controlled, parallel intervention study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Paper Titration Tool and Glooko MIDS (Experimental): Glooko mobile insulin dosing system(MIDS), using the STEP WISE degludec titration algorithm.
  The eligible subjects will be started on insulin degludec (Tresiba® U-200 FlexTouch®). Subjects will use MIDS for insulin degludec titration management. The clinician will configure MIDS Prescription Instruction Form(PIF) using pre-configured Novo Nordisk, Tresiba Protocol Dosing Treatment Plan which is based on the Novo Tresiba degludec Stepwise Program. The Clinician can alter this as appropriate based on medical judgment. Subjects will be started on MIDS and trained on use of Glooko MIDS mobile app. Subjects will get dose adjustment check up on the app and also alert to contact physician if subject experiences hyperglycemia or hypoglycemia.
  Interventions: Device: Glooko Mobile Insulin Dosing System(MIDS)
- Paper Titration tool (No Intervention): Usual care for insulin degludec (Tresiba® U-200 FlexTouch® pens) titration using the STEP WISE degludec titration algorithm.The eligible subjects will be started on insulin degludec(Tresiba® U-200 FlexTouch®).
  Subjects in this group will be provided with a one-page description of the pre-configured Novo Nordisk, Tresiba Protocol Dosing Treatment Plan which is based on the Novo Tresiba degludec Stepwise Program and how to follow it. The Clinician can alter this as appropriate based on medical judgment. This document will also include instructions to contact the HCP if the subject experiences hyperglycemia or hypoglycemia.

INTERVENTIONS:
Device: Glooko Mobile Insulin Dosing System(MIDS) — Mobile Insulin Dosing System (MIDS) for all long acting insulin degludec titration management
  Arms: Paper Titration Tool and Glooko MIDS

SUMMARY:
This is an open label randomized, controlled, parallel intervention study. Group 1 will receive usual care for insulin degludec titration using the STEP WISE degludec titration algorithm Group 2 will receive Glooko mobile insulin dosing system, using the STEP WISE degludec titration algorithm.An estimated n= 240 subjects with type 2 diabetes will be enrolled in order to obtain approximately 200 evaluable subjects who will complete the 16 week study.

DETAILED DESCRIPTION:
This is a prospective randomized controlled two-group parallel design intervention trial. The primary endpoint, change from baseline to week 16 in HbA1c is planned to be tested for superiority of the Glooko Mobile Insulin Dosing System versus standard of care for insulin degludec titration - both with treatment of Tresiba® U-200 FlexTouch®. An estimated n= 240 subjects with type 2 diabetes will be enrolled in order to obtain approximately 200 evaluable subjects who will complete the 16 week study. The subjects, will be already on long-acting insulin or insulin naïve subjects and will be started on long-acting insulin degludec (Tresiba® U-200 FlexTouch®). The subjects will be randomized into one of the two groups: Group 1 will receive standard of care using the STEP WISE degludec titration algorithm for long acting insulin titration. Group 2 will receive standard of care along with treatment facilitated by Glooko mobile insulin dosing system, using the STEP WISE degludec titration algorithm. Major study assessment will be conducted at Baseline (Screening & Visit 1), at a second Visit (Visit 2) after 12 weeks or 3 months and, after 16 weeks or 4 months, a final set of labs, meter download, and subject surveys will be administered (Exit Labs and Meter Download), in addition, any interactions and subsequent care plan changes completed by the HCP during Unscheduled HCP Interactions will be documented. Baseline, Visit 2 and the final screen/Exit Labs visit will include: blood draw, body weight, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has the ability to sign an informed consent form. Prior to randomization patients has signed the informed consent, approved by an Institutional Review Board/Independent Ethics Committee, and provided Health Insurance Portability and Accountability Act authorization (HIPAA) or other privacy authorization prior to any participation in study.
2. Subject 18 and older who has documented type 2 diabetes diagnosis at least 3 months before the screening
3. Subject has HbA1c >/= 7.5% and </=12.5 % measured using a NGSP certified method
4. Subject is initiating basal insulin therapy with insulin degludec or switching to insulin degludec from any basal insulin. The subject may also be on concomitant anti-hyperglycemic agents, including oral hypoglycemic (OAs), non-insulin injectables (e.g. GLP-1) which has been at a stable dose for approx. 3 months, or as determined by the Investigator
5. Subject is a male or non-pregnant, non-lactating female, at least 6 weeks postpartum prior to screening visit. A urine pregnancy test is required for all female subjects unless she is not of childbearing potential, defined as postmenopausal for at least one year prior to screening visit or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy)
6. If female is of childbearing potential, is practicing one of the following methods of birth control (and will continue through the duration of the study):

   1. Condoms, sponge, diaphragm, or intrauterine device;
   2. Oral or parenteral contraceptives for 3 months prior to screening visit;
   3. Vasectomized partner;
   4. Total abstinence from sexual intercourse
7. Subject has a Glooko compatible smart device (smartphone/tablet) with an active data plan or access to Wi-Fi and downloaded at least one mobile application on their phone on their own. If subject does not have a Glooko compatible smart device, a loaner smart device can be provided for the study period.
8. Subject is currently performing self-monitoring of blood glucose(SMBG)

Exclusion Criteria:

1. Subject has had a severe hypoglycemia episode in the last 90 days
2. Subject has type 1 diabetes
3. Subject does not have access to a Glooko compatible smart device (smartphone or tablet)
4. Subject must not be using Glooko or any other electronic application for insulin titration
5. Subject is unable to read and understand English
6. Subject is using short acting or pre-mixed insulin for more than 10 days in the last 3 months
7. Subject is going to initiate short acting insulin prior to the study start
8. Pregnant or breastfeeding women, or the intention of becoming pregnant or not using adequate contraceptive measures
9. Visual impairment resulting in inability to see application.
10. Use of systemic steroids for one week or more in the last 90 days from screening
11. Unable to meet protocol requirements (performing SMBG, administering insulin)
12. Known hypersensitivity / intolerance to insulin degludec or any of its excipients
13. Participant in another clinical study?
14. In the opinion of the PI, if the subject is already on insulin and cannot be properly managed with only long acting insulin (e.g., the introduction of meal time insulin is necessary)
15. Subject has any other condition or event considered exclusionary by the PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | Week 16
  Change in HbA1c at 16 weeks from baseline for all subjects that adhere to treatment.

SECONDARY OUTCOMES:
Change from baseline in HbA1c | Week 12
  Change from baseline in HbA1c
Proportion of synced BG readings < 54 mg/dL | Week 16
  Proportion of synced BG readings < 54 mg/dL
Proportion of synced BG readings < 70 mg/dL | Week 16
  Proportion of synced BG readings < 70 mg/dL
Proportion of synced BG readings >250 mg/dL | Week 16
  Proportion of synced BG readings >250 mg/dL
Proportion of synced BG readings in target range (80-180mg/dL) | Week 16
  Proportion of synced BG readings in target range (80-180mg/dL)
Change in avg BG between first month and last month of study period | Baseline and Week 16
  Change in avg BG between first month and last month of study period
Number of visits to Health Care Professional (HCP) outside of the study visits during study period | Week 16
  Number of visits to Health Care Professional (HCP) outside of the study visits during study period
Number of telephone calls to HCP for insulin titration during study period | Week 16
  Number of telephone calls to HCP for insulin titration during study period
Total insulin degludec dose | Week 12 and Week 16
  Total insulin degludec dose
Change from baseline in Hypoglycemia fear survey- II response | Week 16
  Change from baseline in Hypoglycemia fear survey- II response
Change from baseline in Diabetes Distress Scale (DDS) response | week 16
  Change from baseline in Diabetes Distress Scale (DDS) response
Change from baseline in Diabetes treatment satisfaction questionnaire (DTSQ) response | week 16
  Change from baseline in Diabetes treatment satisfaction questionnaire (DTSQ) response
Number of days with at least one BG test | week 16
  Number of days with at least one BG test
Change from baseline in Body weight | week 16
  Change from baseline in Body weight
Number of Adverse events during study period | week 16
  Number of Adverse events (related/not related)
Number of Serious adverse events during study period | week 16
  Number of Serious Adverse events (related/not related)
Correlation of number of dose adjustment completions to change in HbA1c | week 16
  Correlation of number of dose adjustment completions to change in HbA1c
Number of subjects that have attained an avg fasting blood glucose target range for at least three of last five titration cycles of study period during trial | week 16
  For MIDS arm only
Number of dose adjustments to first reach avg FBG target range during study period | week 16
  For MIDS arm only
Total insulin degludec dose for subjects who reached avg FBG target at last dose checkup. | week 16
  For MIDS arm only
Frequency of FBG tests during study period | week 16
  For MIDS arm only
Proportion of accepted MIDS recommended insulin degludec doses | week 16
  For MIDS arm only

CONTACTS AND LOCATIONS:
Overall Officials: Michael Greenfield, MD, Study Director — Glooko
Locations (1):
- Scripps Whittier Diabetes Institute, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] IDF 2015 Atlas: http://www.diabetesatlas.org/resources/2015-atlas. html
- [Background] Centers for Disease Control and Prevention (CDC), Diabetes Public Health Resource. Number (in Millions) of Adults with Diabetes by Diabetes Medication Status, United States, 1997-2011: http://www. cdc.gov/diabetes/statistics/meduse/fig1.htm
- [Background] Ali MK, McKeever Bullard K, Imperatore G, Barker L, Gregg EW; Centers for Disease Control and Prevention (CDC). Characteristics associated with poor glycemic control among adults with self-reported diagnosed diabetes--National Health and Nutrition Examination Survey, United States, 2007-2010. MMWR Suppl. 2012 Jun 15;61(2):32-7. PMID 22695461
- [Background] Donnelly LA, Morris AD, Evans JM; DARTS/MEMO collaboration. Adherence to insulin and its association with glycaemic control in patients with type 2 diabetes. QJM. 2007 Jun;100(6):345-50. doi: 10.1093/qjmed/hcm031. Epub 2007 May 15. PMID 17504861
- [Background] Peyrot M, Rubin RR, Kruger DF, Travis LB. Correlates of insulin injection omission. Diabetes Care. 2010 Feb;33(2):240-5. doi: 10.2337/dc09-1348. PMID 20103556
- [Background] Yurgin NR, Boye KS, Dilla T, Surinach NL, Llach XB. Physician and patient management of type 2 diabetes and factors related to glycemic control in Spain. Patient Prefer Adherence. 2008 Feb 2;2:87-95. PMID 19920948
- [Background] Peyrot M, Barnett AH, Meneghini LF, Schumm-Draeger PM. Insulin adherence behaviours and barriers in the multinational Global Attitudes of Patients and Physicians in Insulin Therapy study. Diabet Med. 2012 May;29(5):682-9. doi: 10.1111/j.1464-5491.2012.03605.x. PMID 22313123
- [Background] Cramer JA, Pugh MJ. The influence of insulin use on glycemic control: How well do adults follow prescriptions for insulin? Diabetes Care. 2005 Jan;28(1):78-83. doi: 10.2337/diacare.28.1.78. PMID 15616237
- [Background] Balkrishnan R, Rajagopalan R, Camacho FT, Huston SA, Murray FT, Anderson RT. Predictors of medication adherence and associated health care costs in an older population with type 2 diabetes mellitus: a longitudinal cohort study. Clin Ther. 2003 Nov;25(11):2958-71. doi: 10.1016/s0149-2918(03)80347-8. PMID 14693318
- [Background] Chandran A, Bonafede MK, Nigam S, Saltiel-Berzin R, Hirsch LJ, Lahue BJ. Adherence to Insulin Pen Therapy Is Associated with Reduction in Healthcare Costs Among Patients with Type 2 Diabetes Mellitus. Am Health Drug Benefits. 2015 May;8(3):148-58. PMID 26085903
- [Background] Cuddihy RM, Philis-Tsimikas A, Nazeri A. Type 2 diabetes care and insulin intensification: is a more multidisciplinary approach needed? Results from the MODIFY survey. Diabetes Educ. 2011 Jan-Feb;37(1):111-23. doi: 10.1177/0145721710388426. Epub 2010 Dec 3. PMID 21131599
- [Background] Nichols GA, Koo YH, Shah SN. Delay of insulin addition to oral combination therapy despite inadequate glycemic control: delay of insulin therapy. J Gen Intern Med. 2007 Apr;22(4):453-8. doi: 10.1007/s11606-007-0139-y. PMID 17372792
- [Background] Peyrot M, Rubin RR, Lauritzen T, Skovlund SE, Snoek FJ, Matthews DR, Landgraf R, Kleinebreil L; International DAWN Advisory Panel. Resistance to insulin therapy among patients and providers: results of the cross-national Diabetes Attitudes, Wishes, and Needs (DAWN) study. Diabetes Care. 2005 Nov;28(11):2673-9. doi: 10.2337/diacare.28.11.2673. PMID 16249538
- [Background] Strain WD, Bluher M, Paldanius P. Clinical inertia in individualising care for diabetes: is there time to do more in type 2 diabetes? Diabetes Ther. 2014 Dec;5(2):347-54. doi: 10.1007/s13300-014-0077-8. Epub 2014 Aug 12. PMID 25113408
- [Background] Hayes RP, Fitzgerald JT, Jacober SJ. Primary care physician beliefs about insulin initiation in patients with type 2 diabetes. Int J Clin Pract. 2008 Jun;62(6):860-8. doi: 10.1111/j.1742-1241.2008.01742.x. Epub 2008 Apr 3. PMID 18393965
- [Background] Ratanawongsa N, Crosson JC, Schillinger D, Karter AJ, Saha CK, Marrero DG. Getting under the skin of clinical inertia in insulin initiation: the Translating Research Into Action for Diabetes (TRIAD) Insulin Starts Project. Diabetes Educ. 2012 Jan-Feb;38(1):94-100. doi: 10.1177/0145721711432649. Epub 2012 Jan 5. PMID 22222513
- [Background] Karter AJ, Subramanian U, Saha C, Crosson JC, Parker MM, Swain BE, Moffet HH, Marrero DG. Barriers to insulin initiation: the translating research into action for diabetes insulin starts project. Diabetes Care. 2010 Apr;33(4):733-5. doi: 10.2337/dc09-1184. Epub 2010 Jan 19. PMID 20086256
- [Background] Strain WD, Cos X, Hirst M, Vencio S, Mohan V, Voko Z, Yabe D, Bluher M, Paldanius PM. Time to do more: addressing clinical inertia in the management of type 2 diabetes mellitus. Diabetes Res Clin Pract. 2014 Sep;105(3):302-12. doi: 10.1016/j.diabres.2014.05.005. Epub 2014 May 27. PMID 24956964
- [Background] Sorli C, Heile MK. Identifying and meeting the challenges of insulin therapy in type 2 diabetes. J Multidiscip Healthc. 2014 Jul 2;7:267-82. doi: 10.2147/JMDH.S64084. eCollection 2014. PMID 25061317
- [Background] Blonde L, Merilainen M, Karwe V, Raskin P; TITRATE Study Group. Patient-directed titration for achieving glycaemic goals using a once-daily basal insulin analogue: an assessment of two different fasting plasma glucose targets - the TITRATE study. Diabetes Obes Metab. 2009 Jun;11(6):623-31. doi: 10.1111/j.1463-1326.2009.01060.x. PMID 19515182
- [Background] Meneghini L, Koenen C, Weng W, Selam JL. The usage of a simplified self-titration dosing guideline (303 Algorithm) for insulin detemir in patients with type 2 diabetes--results of the randomized, controlled PREDICTIVE 303 study. Diabetes Obes Metab. 2007 Nov;9(6):902-13. doi: 10.1111/j.1463-1326.2007.00804.x. PMID 17924873
- [Background] Davies M, Lavalle-Gonzalez F, Storms F, Gomis R; AT.LANTUS Study Group. Initiation of insulin glargine therapy in type 2 diabetes subjects suboptimally controlled on oral antidiabetic agents: results from the AT.LANTUS trial. Diabetes Obes Metab. 2008 May;10(5):387-99. doi: 10.1111/j.1463-1326.2008.00873.x. Epub 2008 Mar 18. PMID 18355327
- [Background] Pew Research Center: http://www.pewinternet.org/2015/10/29/ technology-device-ownership-2015/ (accessed May 18, 2016)
- [Background] Walker RJ, Smalls BL, Hernandez-Tejada MA, Campbell JA, Egede LE. Effect of diabetes self-efficacy on glycemic control, medication adherence, self-care behaviors, and quality of life in a predominantly low-income, minority population. Ethn Dis. 2014 Summer;24(3):349-55. PMID 25065078
- [Background] Hou C, Carter B, Hewitt J, Francisa T, Mayor S. Do Mobile Phone Applications Improve Glycemic Control (HbA1c) in the Self-management of Diabetes? A Systematic Review, Meta-analysis, and GRADE of 14 Randomized Trials. Diabetes Care. 2016 Nov;39(11):2089-2095. doi: 10.2337/dc16-0346. PMID 27926892
- See also: Pew Research Center(accessed May 18, 2016) — http://www.pewinternet.org/2015/10/29/technology-device-ownership-2015/